CLINICAL TRIAL: NCT01998087
Title: The Effect of Written Information and Support Phone Calls for First Time Mothers on Breastfeeding Rates: A Randomized Controlled Trial
Brief Title: Proactive Breastfeeding Support in First Time Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Irena Zakarija-Grkovic, Lecturer/researcher, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2181-198-03-04-13-0027
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Breastfeeding
Keywords: Exclusive breastfeeding; Breastfeeding; Proactive breastfeeding support; Telephone breastfeeding support; Infant feeding attitudes; Breastfeeding self-efficacy; Breastfeeding difficulties
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breastfeeding support (Experimental): A breastfeeding brochure will be distributed to expectant mothers from 20 weeks gestation during their regular antenatal visit. This will be followed 2 weeks later by a phone call offering clarification/explanation of the brochure. Three standardized phone calls, offering breastfeeding support, will be conducted at 2,6 and 10 weeks following birth of the baby.
  Interventions: Behavioral: Breastfeeding support
- General Support (Active Comparator): The active control group of mothers will receive a brochure in pregnancy covering general pregnancy and parenting issues and follow-up phone calls but breastfeeding issues will not be specifically addressed. If a mother raises any breastfeeding issue she will be referred to appropriate support.
  Interventions: Behavioral: Breastfeeding support
- Standard Care (No Intervention): This group will receive standard antenatal care provided by their chosen gynaecologist and obstetrician, consisting of regular antenatal visits. No written materials or telephone calls are routinely provided to pregnant women in Croatia.

INTERVENTIONS:
Behavioral: Breastfeeding support — A breastfeeding brochure will be distributed to expectant mothers from 20 weeks gestation during their regular antenatal visit. This will be followed 2 weeks later by a phone call offering clarification/explanation of the brochure. Three phone calls, offering breastfeeding support, will be conducted at 2,6 and 10 weeks following the birth of the baby.
  Arms: Breastfeeding support; General Support

SUMMARY:
In Croatia, between 95% and 99% of mothers initiate breastfeeding, but by 3 months a third have stopped, and by six months only half are still providing any human milk for their babies. Exclusive breastfeeding rates are even lower, with only about 9% of Croatian mothers exclusively breastfeeding at 6 months, despite the WHO recommendation of 6 months of exclusive breastfeeding. Currently, in Croatia, no breastfeeding information or other pregnancy and parenting related written information is routinely provided to expectant couples. In our study we would like to find out whether providing written breastfeeding information in pregnancy and breastfeeding focused support phone calls during pregnancy and after the birth of the baby result in better outcomes than providing general pregnancy/parenting information and support phone calls. This will be tested by randomising women, attending their primary health care provider for routine antenatal visits between 20 and 32 weeks, to an intervention focused on promoting and supporting breastfeeding, to an intervention focused on general pregnancy and parenting issues, and to a non-intervention control group. Women will be followed-up for 6 months after the birth of their baby and data will be collected at 3 and 6 months on breastfeeding rates, breastfeeding self-efficacy, breastfeeding difficulties, social support and attitudes toward infant feeding.

ELIGIBILITY:
Inclusion Criteria:

* expectant women, between 20 and 32 weeks gestation, attending any of 6 pre- determined antenatal clinics
* primigravidae
* singleton pregnancy
* can read and write Croatian
* resides in Croatia or plans to stay in Croatia at least 12 months following the birth

Exclusion Criteria:

* multigravidae
* women expecting twins/multiples
* refuses to participate
* inability to communicate in Croatian by phone
* planning to leave the County of Split Dalmatia within a year of giving birth
* severe maternal psychiatric or medical problems

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 3 months

SECONDARY OUTCOMES:
Any breastfeeding | 3 & 6 months

OTHER OUTCOMES:
Maternal attitudes toward infant feeding | Before (at recruitment) and after (at 3 months)
  Validated Iowa Infant Feeding Attitude Scale to be used.
Breastfeeding self-efficacy scale | At 3 months post birth
  Validated tool measuring a mother's confidence in her ability to breastfeed
Breastfeeding difficulties | At 3 months postbirth

CONTACTS AND LOCATIONS:
Overall Officials: Irena Zakarija-Grkovic, MD, PhD, Principal Investigator — University of Split
Locations (1):
- Cito Obstetrics and Gynaecology Clinic, Split, Outside AUS, Croatia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Puharic D, Malicki M, Borovac JA, Sparac V, Poljak B, Aracic N, Marinovic N, Luetic N, Zakarija-Grkovic I. The effect of a combined intervention on exclusive breastfeeding in primiparas: A randomised controlled trial. Matern Child Nutr. 2020 Jul;16(3):e12948. doi: 10.1111/mcn.12948. Epub 2020 Jan 13. PMID 31943761